CLINICAL TRIAL: NCT01445951
Title: A Phase 3, Multicenter, Open-label, Randomized, Forced-titration Clinical Trial Evaluating the Efficacy and Safety of Technosphere® Insulin Inhalation Powder in Combination With a Basal Insulin Versus Insulin Aspart in Combination With a Basal Insulin in Subjects With Type 1 Diabetes Mellitus Over a 24-week Treatment Period
Brief Title: Clinical Trial Evaluating Technosphere® Insulin Versus Insulin Aspart in Subjects With Type 1 Diabetes Mellitus Over a 24-week Treatment Period
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-171
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Technosphere® Insulin with MedTone C Inhaler (Experimental): Subjects will receive TI with the MedToneC inhaler and remain on the basal insulin they were taking prior to study entry
  Interventions: Drug: Technosphere® Insulin with MedTone C Inhaler
- Aspart Group (Active Comparator): Subjects will receive insulin aspart and remain on the basal insulin they were taking prior to study entry
  Interventions: Drug: Insulin Aspart in combination with a basal insulin
- Technosphere ® Insulin-Gen2 Group (Experimental): Subject will receive Technosphere Insulin with Gen2 Inhaler and remain on the basal insulin they were taking prior to study entry
  Interventions: Drug: Technosphere ®Insulin with Gen2 Inhaler

INTERVENTIONS:
Drug: Technosphere® Insulin with MedTone C Inhaler — Inhalation Powder and injectable insulin
  Arms: Technosphere® Insulin with MedTone C Inhaler
Drug: Technosphere ®Insulin with Gen2 Inhaler — Inhalation Powder and injectable insulin
  Arms: Technosphere ® Insulin-Gen2 Group
Drug: Insulin Aspart in combination with a basal insulin — Injectable insulin
  Arms: Aspart Group

SUMMARY:
Open-label, randomized, forced-titration clinical trial evaluating the efficacy and safety of TI Inhalation Power in combination with a basal insulin versus insulin aspart in combination with a basal insulin

DETAILED DESCRIPTION:
Phase 3 clinical trial designed to examine the efficacy and safety of inhaled prandial TI Inhalation Power in combination with basal insulin versus insulin aspart in combination with basal insulin in subjects with type 1 diabetes who are suboptimally controlled with their current insulin regimens. This trial will employ a variety of methods to intensively manage these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women = 18 years of age
* Clinical diagnosis of type 1 diabetes mellitus for at least 12 months
* Body mass index (BMI) = 38 kg/m2
* Stable dose of basal/bolus insulin therapy for at least 3 months with an FPG consistently < 220 mg/dL:
* HbA1c = 7.5% and = 10.0%
* Fasting C-peptide = 0.30 pmol/mL
* Subject willingness to not use CGM during the entire course of the trial
* Nonsmoking (includes cigarettes, cigars, pipes, and chewing tobacco) for the preceding 6 months
* Negative urine cotinine test, defined as = 100 ng/mL
* Lung function tests: • Forced expiratory volume in 1 second (FEV1) = 70% Third National Health and Nutrition Examination Survey (NHANES III) predicted
* Written informed consent

Exclusion Criteria:

* Total daily insulin dose = 2 IU/kg/day. History of insulin pump use within 3 months of Screening or use of continuous glucose monitoring within 6 weeks of Screening
* History of inhaled insulin use in the previous 6 months
* Two or more unexplained severe hypoglycemic episodes within 3 months of Screening or an episode of severe hypoglycemia between Visit 1 and Visit 2. Unexplained refers to episodes of severe hypoglycemia that are not related to a dosing error, lack of or a change in meal size, or related to additional/unanticipated exercise
* Any hospitalization or emergency room visit due to poor diabetic control within 6 months of Screening, or hospitalization or emergency room visit due to poor diabetic control between Visit 1 and Visit 2
* Allergy or known hypersensitivity to insulin or to any of the drugs to be used in the study, or a history of hypersensitivity to TI Inhalation Powder or to drugs with a similar chemical structure
* History of recent blood transfusions (within previous 3 months), hemoglobinopathies, or any other conditions that affect HbA1c measurements.
* History of COPD, asthma, or any other clinically important pulmonary disease (eg, pulmonary fibrosis), or use of any medications for these conditions
* Any clinically significant radiological findings on screening chest x-ray
* Active respiratory infection within 30 days before Screening (subject may return after 30 days from resolution for rescreening)
* Major organ system diseases, including: ? Seizure disorder; systemic autoimmune or collagen vascular disease requiring previous or current treatment with systemic corticosteroids, cytotoxic drugs, or penicillamine; cancer (other than excised cutaneous basal cell carcinoma) or any history of lung neoplasms
* Current or previous chemotherapy or radiation therapy that may result in pulmonary toxicity; use of medications for weight loss (eg, sibutramine, orlistat) within 12 weeks of Screening; treatment with amiodarone within 12 weeks of Screening
* Clinically significant abnormalities on screening laboratory evaluation or chest x-ray
* Severe complications of diabetes, in the opinion of the PI, including symptomatic autonomic neuropathy; disabling peripheral neuropathy; active proliferative retinopathy; nephropathy with renal failure, renal transplant, or dialysis; nontraumatic amputations due to gangrene; or vascular claudication
* Women who are pregnant, lactating, or planning to become pregnant during the clinical study period; women of childbearing potential (defined as premenopausal and not surgically sterilized or postmenopausal for fewer than 2 years) not practicing adequate birth control. Adequate birth control is defined as using oral, percutaneous, or transdermal contraceptives; condoms and diaphragms (double barrier) with a spermicide; or intrauterine devices. Postmenopausal for this study includes amenorrhea f
* Current drug or alcohol abuse or a history of drug or alcohol abuse that, in the opinion of the PI, would make the subject an unsuitable candidate for participation in the study
* Exposure to any investigational medications or devices within the previous 30 days before study entry
* Unable to read or write, or unlikely to comprehend and follow the study protocol procedures; lack of compliance with medication or procedures that, in the PI's opinion, may affect the study data or subject safety and that precludes the subject from participation in the study; or any other concurrent medical or major psychiatric condition that, in the opinion of the PI, makes the subject unsuitable for the clinical study or could limit the validity of the informed consent or impair the subject'

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (53):
  - Burlingame, California
  - Escondido, California
  - Huntington Beach, California
  - La Jolla, California
  - La Mesa, California
  - Long Beach, California
  - Los Angeles, California
  - Los Gatos, California
  - San Mateo, California
  - Santa Barbara, California
  - Tustin, California
  - Aurora, Colorado
  - Hialeah, Florida
  - Hollywood, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Palm Harbor, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Dunwoody, Georgia
  - Lawrenceville, Georgia
  - Roswell, Georgia
  - Chicago, Illinois
  - Vincennes, Indiana
  - Des Moines, Iowa
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Edina, Minnesota
  - City of Saint Peters, Missouri
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Paramus, New Jersey
  - Albuquerque, New Mexico
  - Flushing, New York
  - New Hyde Park, New York
  - New York, New York
  - Asheville, North Carolina
  - Greenville, North Carolina
  - Morehead City, North Carolina
  - Portland, Oregon
  - Greer, South Carolina
  - Bartlett, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Federal Way, Washington
  - Renton, Washington
  - Wenatchee, Washington
- Brazil (2):
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Russia (7):
  - Saint Petersburg, Russia
  - Kemerovo, RUS
  - Moscow, RUS
  - Petrozavodsk, RUS
  - Saint Petersburg, RUS
  - Smolensk, RUS
  - Yaroslavl, RUS
- Ukraine (7):
  - Dnipropetrovsk, UKR
  - Donetsk, UKR
  - Kharkiv, UKR
  - Kiev, UKR
  - Kyiv, UKR
  - Odesa, UKR
  - Vinnytsia, UKR

REFERENCES:
- [Derived] Seaquist ER, Blonde L, McGill JB, Heller SR, Kendall DM, Bumpass JB, Pompilio FM, Grant ML. Hypoglycaemia is reduced with use of inhaled Technosphere(R) Insulin relative to insulin aspart in type 1 diabetes mellitus. Diabet Med. 2020 May;37(5):752-759. doi: 10.1111/dme.14202. Epub 2019 Dec 19. PMID 31811662
- [Derived] Bode BW, McGill JB, Lorber DL, Gross JL, Chang PC, Bregman DB; Affinity 1 Study Group. Inhaled Technosphere Insulin Compared With Injected Prandial Insulin in Type 1 Diabetes: A Randomized 24-Week Trial. Diabetes Care. 2015 Dec;38(12):2266-73. doi: 10.2337/dc15-0075. Epub 2015 Jul 15. PMID 26180109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient enrolled Sept 2011. Multi-national trial conducted in US, Russia, Ukraine and Brazil.
Pre-assignment Details: 3 week Screening Period prior to run-in (basal insulin optimization period). 1401 Screened / 621 Eligible of which 614 entered the run-in period. 538 met randomization criteria at end of run-in of which 518 were randomized.
Groups:
- Technosphere Insulin-Gen2 + Basal Insulin: Technosphere Insulin delivered via the Gen2 Inhaler plus subcutaneous basal insulin, doses individualized for each patient
- Technosphere Insulin-MedTone + Basal Insulin: Technosphere Insulin delivered via the MedTone C Inhaler plus subcutaneous basal insulin, doses individualized for each patient
- Insulin Aspart + Basal Insulin: Subcutaneous insulin aspart plus subcutaneous basal insulin, doses individualized for each patient
Period: Overall Study
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Started | 174 | 174 | 170
Completed | 130 | 138 | 151
Not Completed | 44 | 36 | 19
Not completed — Adverse Event | 16 | 9 | 0
Not completed — Protocol Violation | 2 | 2 | 2
Not completed — Withdrawal by Subject | 21 | 16 | 8
Not completed — Physician Decision | 3 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 4
Not completed — Pregnancy | 0 | 1 | 4
Not completed — Death | 0 | 0 | 1
Not completed — Non-compliance with study drug | 1 | 2 | 0
Not completed — Non-compliance with protocol | 0 | 1 | 0
Not completed — Sponsor decision - subject travel | 0 | 1 | 0
Not completed — Cough | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin | Total
Number analyzed (Participants) | 174 | 174 | 170 | 518
Age, Customized [Number; unit: participants]
  18-30 years | 56 | 48 | 46 | 150
  31-49 years | 93 | 84 | 88 | 265
  50-64 years | 18 | 33 | 28 | 79
  >= 65 years | 7 | 9 | 8 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 94 | 96 | 287
  Male | 77 | 80 | 74 | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 22 | 18 | 57
  Not Hispanic or Latino | 157 | 152 | 152 | 461
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 8 | 5 | 3 | 16
  White | 164 | 167 | 166 | 497
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 71 | 69 | 67 | 207
  Brazil | 14 | 15 | 13 | 42
  Ukraine | 44 | 38 | 38 | 120
  Russian Federation | 45 | 52 | 52 | 149
Duration of Diabetes [Mean (Full Range); unit: years] | 16.0 [1.1 to 57.3] | 17.7 [1.1 to 49.5] | 16.7 [1.0 to 42.2] | 16.8 [1.0 to 57.3]
Weight [Mean (Full Range); unit: kg] | 75.7 [41.7 to 129.4] | 76.8 [47.6 to 124.0] | 72.6 [46.6 to 120.2] | 75.1 [41.7 to 129.4]
BMI [Mean (Full Range); unit: kg/m^2] | 26.0 [16.6 to 38.6] | 26.2 [18.1 to 36.4] | 25.4 [17.4 to 37.2] | 25.9 [16.6 to 38.6]
Fasting Plasma Glucose [Mean (Full Range); unit: mg/dL] | 155.0 [21.0 to 403.0] | 144.3 [43.0 to 358.0] | 151.2 [23.0 to 375.0] | 150.2 [21.0 to 403.0]
HbA1c [Mean (Full Range); unit: Percent of hemoglobin] | 7.98 [6.20 to 10.60] | 8.00 [6.10 to 10.20] | 7.88 [5.80 to 10.10] | 7.95 [5.80 to 10.60]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in HbA1c
Description: Effect of treatment as measured by change from baseline in glycated hemoglobin (HbA1c). Primary treatment difference is TI-Gen2 vs. Insulin Aspart at Week 24
Time Frame: Baseline to Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Percent of hemoglobin
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 174 | 174 | 170
Percent of hemoglobin | -0.21 (0.062) | -0.29 (0.061) | -0.40 (0.060)
Statistical Analysis 1: Comparison: Technosphere Insulin-Gen2 + Basal Insulin vs Insulin Aspart + Basal Insulin; MMRM (mixed model repeated measures) model with auto-regression (1): HbA1c = Baseline HbA1c + region + basal insulin stratum + visit + treatment + (visit*treatment); Test type: Non-Inferiority or Equivalence — Non-inferiority with 0.4 margin; Mean Difference (Net) = 0.19, 95% CI 2-sided [0.02 to 0.36], Standard Error of Mean 0.086

2. Secondary Outcome: FEV1 Change From Baseline to Week 24
Description: Forced Expiratory Volume in 1 second - change from baseline to week 24
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 174 | 173 | 171
Liters | -0.07 (0.012) | -0.08 (0.012) | -0.04 (0.011)
Statistical Analysis 1: Comparison: Technosphere Insulin-Gen2 + Basal Insulin vs Technosphere Insulin-MedTone + Basal Insulin; Test type: Superiority or Other; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.02 to 0.04], Standard Error of Mean 0.016 — Mixed Model Repeated Measure (MMRM): FEV1 = Baseline FEV1 + Age + Gender + Race + Baseline Height + Visit + Treatment + (Visit*Treatment)

3. Secondary Outcome: FPG Change From Baseline to Week 24
Description: Comparison of mean change from Baseline to Week 24 visit in fasting plasma glucose (FPG) levels (central laboratory results)
Time Frame: Baseline to Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 174 | 174 | 170
mg/dL | -25.27 (7.62) | 7.15 (7.53) | 10.15 (7.40)
Statistical Analysis 1: Comparison: Technosphere Insulin-Gen2 + Basal Insulin vs Insulin Aspart + Basal Insulin; Test type: Superiority or Other; Mean Difference (Net) = -35.42, 95% CI 2-sided [-56.25 to -14.59], Standard Error of Mean 10.622 — MMRM: FPG = Baseline FPG + Region + Basal insulin stratum + Visit + Treatment + (Visit*Treatment)

4. Secondary Outcome: Mean 7-point Glucose Baseline Values
Description: Mean 7-point glucose at baseline
Time Frame: Baseline
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 174 | 174 | 170
mg/dL
  Before breakfast | 154.1 (38.85) | 151.8 (40.32) | 147.0 (39.09)
  After breakfast | 173.3 (48.77) | 173.5 (48.36) | 162.6 (49.50)
  Before lunch | 158.0 (47.39) | 156.6 (42.91) | 142.3 (37.86)
  After lunch | 169.5 (52.25) | 169.7 (49.23) | 157.6 (48.08)
  Before dinner | 169.9 (47.12) | 168.1 (45.24) | 154.0 (46.53)
  After dinner | 176.2 (51.55) | 177.0 (53.17) | 158.5 (47.64)
  Bedtime | 178.3 (51.38) | 175.1 (43.99) | 164.4 (49.97)

5. Secondary Outcome: Mean 7-point Glucose Week 24 Values
Time Frame: Week 24
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 174 | 174 | 170
mg/dL
  Before breakfast | 148.2 (40.64) | 147.9 (43.17) | 155.3 (48.44)
  After breakfast | 169.7 (67.53) | 164.1 (60.97) | 163.0 (58.00)
  Before lunch | 168.2 (56.93) | 165.9 (59.95) | 149.1 (50.58)
  After lunch | 173.7 (57.09) | 163.1 (50.92) | 158.2 (50.04)
  Before dinner | 177.8 (59.96) | 177.3 (56.71) | 156.8 (48.30)
  After dinner | 180.8 (63.50) | 168.2 (60.77) | 157.8 (52.62)
  Bedtime | 185.2 (62.36) | 185.6 (54.96) | 175.4 (57.37)

6. Secondary Outcome: Change in Body Weight From Baseline to Week 24
Description: Change in body weight from Baseline to Week 24
Time Frame: Baseline to Week 24
Population: Full analysis set (subjects with data available at Baseline and at Week 24)
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 132 | 140 | 153
kg | -0.39 (0.438) | -0.19 (0.428) | 0.93 (0.441)
Statistical Analysis 1: Comparison: Technosphere Insulin-Gen2 + Basal Insulin vs Insulin Aspart + Basal Insulin; Test type: Superiority or Other; p = 0.0102, ANCOVA; ANCOVA: Weight change from baseline = Baseline weight + Change from baseline in HbA1c + Region + Basal insulin stratum + Treatment; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-2.33 to -0.31], Standard Error of Mean 0.512 — ANCOVA: Weight change from baseline = Baseline weight + Change from baseline in HbA1c + Region + Basal insulin stratum + Treatment
Statistical Analysis 2: Comparison: Technosphere Insulin-Gen2 + Basal Insulin; Within treatment analysis of change from Baseline comparing if change was different from zero; Test type: Superiority or Other; p = 0.4955, t-test, 2 sided
Statistical Analysis 3: Comparison: Technosphere Insulin-MedTone + Basal Insulin; Within treatment analysis of change from Baseline comparing if change was different from zero; Test type: Superiority or Other; p = 0.6807, t-test, 2 sided
Statistical Analysis 4: Comparison: Insulin Aspart + Basal Insulin; Within treatment analysis of change from Baseline comparing if change was different from zero; Test type: Superiority or Other; p = 0.0079, t-test, 2 sided

7. Other Pre Specified Outcome: Incidence of Total Hypoglycemia
Description: Hypoglycemia, defined as blood glucose <= 70 mg/dL or in absence of blood glucose, symptoms that are resolved by the administration of carbohydrates.
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 174 | 173 | 171
percentage of participants | 96.0 | 96.0 | 99.4

8. Other Pre Specified Outcome: Incidence of Severe Hypoglycemia
Description: Severe Hypoglycemia defined as: Requiring 3rd party assistance.
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 174 | 173 | 171
percentage of participants | 18.4 | 21.4 | 29.2
Statistical Analysis 1: Comparison: Technosphere Insulin-Gen2 + Basal Insulin vs Insulin Aspart + Basal Insulin; Test type: Superiority or Other; p = 0.0156, Regression, Logistic; Logistic model with affects for Region, Basal insulin stratum, and Treatment; Odds Ratio (OR) = 0.5328, 95% CI 2-sided [0.3198 to 0.8877]

9. Other Pre Specified Outcome: Total Hypoglycemia Event Rate
Description: Number of Hypoglycemic Events/Total Subject Exposure Time (in months)
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Number; unit: Events/Subject-Month
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 174 | 173 | 171
Events/Subject-Month | 9.80 | 10.30 | 13.97
Statistical Analysis 1: Comparison: Technosphere Insulin-Gen2 + Basal Insulin vs Insulin Aspart + Basal Insulin; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression; Model: Region + Basal Insulin Stratum + Treatment + Exposure Time

10. Other Pre Specified Outcome: Severe Hypoglycemia Event Rate
Description: Number of Severe Hypoglycemic Events/Total Subject Exposure Time (in months)
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Number; unit: Events/Subject-Month
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 174 | 173 | 171
Events/Subject-Month | 8.05 | 9.99 | 14.45
Statistical Analysis 1: Comparison: Technosphere Insulin-Gen2 + Basal Insulin vs Insulin Aspart + Basal Insulin; Test type: Superiority or Other; p = 0.1022, Negative Binomial Regression; Model: Region + Basal Insulin Stratum + Treatment + Exposure Time

11. Secondary Outcome: Proportion of Responders Achieving HbA1c <= 7.0%
Description: Efficacy as measured in proportion of subjects achieving HbA1c < or = to 7.0%
Time Frame: Week 24
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Technosphere Insulin-Gen2 + Basal Insulin | Technosphere Insulin-MedTone + Basal Insulin | Insulin Aspart + Basal Insulin
Number analyzed (Participants) | 131 | 138 | 150
percentage of participants | 18.3 | 21.7 | 30.7
Statistical Analysis 1: Comparison: Technosphere Insulin-Gen2 + Basal Insulin vs Insulin Aspart + Basal Insulin; Test type: Superiority or Other; p = 0.0158, Regression, Logistic; Model: Treatment + Basal insulin stratum + Region + Baseline HbA1c; Odds Ratio (OR) = 0.449, 95% CI 2-sided [0.23 to 0.86] — Gen2 in the numerator, Aspart in the denominator

ADVERSE EVENTS:
Time Frame: Baseline to Week 24
Description: Adverse Events (AE) are summarized according to how subjects were treated, not randomized. One subject that was randomized to the Technosphere Insulin-MedTone + Basal Insulin arm was treated with Insulin aspart + Basal Insulin throughout the trial.
Arm/Group | Technosphere ® Insulin-Gen2 Group | Technosphere® Insulin With MedTone C Inhaler | Aspart Group
Serious Adverse Events (participants affected / at risk) | 5/174 | 9/173 | 7/171
Other Adverse Events (participants affected / at risk) | 81/174 | 74/173 | 50/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Technosphere ® Insulin-Gen2 Group (N=174) | Technosphere® Insulin With MedTone C Inhaler (N=173) | Aspart Group (N=171)
Chest Discomfort (General disorders) | 0 | 1 | 0
Drowning (General disorders) | 0 | 0 | 1
Cytomegalovirus Infection (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypoglycaemic Unconsciousness (Nervous system disorders) | 1 | 4 | 2
Hypoglycaemic Seizure (Nervous system disorders) | 1 | 1 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1
Cervical Polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Technosphere ® Insulin-Gen2 Group (N=174) | Technosphere® Insulin With MedTone C Inhaler (N=173) | Aspart Group (N=171)
Cough (Respiratory, thoracic and mediastinal disorders) | 55 | 39 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 14 | 16 | 12
Headache (Nervous system disorders) | 7 | 5 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 1 | 4
Nasopharyngitis (Infections and infestations) | 5 | 13 | 12
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 3
Influenza (Infections and infestations) | 2 | 9 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3 | 5
Urinary Tract Infection (Infections and infestations) | 1 | 6 | 3
Nausea (Gastrointestinal disorders) | 1 | 5 | 6
Blood Creatine Phosphokinase Increase (Investigations) | 0 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.